CLINICAL TRIAL: NCT01553214
Title: Collection of Granulocytes by Apheresis of Healthy Donors Stimulated With Filgrastim (G-CSF) and Dexamethasone
Brief Title: Improving White Blood Cell Collection From Healthy Donors
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 120096; 12-CC-0096
Record Dates: First submitted 2012-03-10; First posted 2012-03-14 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-23

CONDITIONS: Allogeneic Granulocyte Donation
Keywords: Neutrophils; Infection; Granulocytapheresis; Mobilization; Transfusion; Healthy Volunteer; HV
MeSH Terms: conditions — Infections | interventions — Filgrastim; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Donors (Other): volunteer healthy donors willing to receive G-CSF and dexamethasone and undergo leukapheresis
  Interventions: Drug: Filgrastim; Drug: Dexamethasone

INTERVENTIONS:
Drug: Filgrastim — Donors shall receive G-CSF 480 mcg as a single 1.6-mL subcutaneous injection 12 to 24 hours prior to donation.
Drug: Dexamethasone — Donors shall ingest dexamethasone 8 mg (two 4-mg tablets) orally 12 hours prior to donation.

SUMMARY:
Background:

- White blood cells called granulocytes help the body fight infection. People who have had chemotherapy or bone marrow transplants may have very low numbers of these cells. Transfusions of these cells can help improve the body's ability to fight infection. However, most of the cells are located in the bone marrow or spleen, and are hard to collect from healthy donors. Two drugs, filgrastim and dexamethasone, can help move the cells to the bloodstream to be collected by apheresis. Researchers want to study the best ways to collect these white blood cells. They also want to monitor the effects of the injections and donations on the volunteer donors.

Objectives:

- To improve the amount and quality of granulocytes (white blood cells) collected by apheresis for donation.

Eligibility:

- Healthy volunteers between 18 and 75 years of age.

Design:

* Participants will be screened with a physical exam and medical history. Initial blood tests will be done to check for eligibility.
* Participants will donate granulocytes by apheresis a maximum of 12 times in 1 year. Donations will not usually be requested more often than every 4 weeks. Donors will be allowed to decline participation at any time.
* Participants will have one injection of filgrastim 12 to 24 hours before donation. They will also have two tablets of dexamethasone 12 hours before donation.
* White blood cells will be collected through apheresis. The apheresis will last about 2 hours.
* Participants will be eligible to donate until they reach their 76th birthday....

DETAILED DESCRIPTION:
Bacterial and fungal infections in neutropenic patients or in patients with inherited disorders of neutrophil function continue to cause substantial morbidity and mortality. In particular, fungal infections are an increasingly important cause of death in patients receiving aggressive chemotherapy, in patients undergoing hematopoietic stem cell transplantation (HSCT), in patients with chronic granulomatous disease, and in patients with bone marrow failure syndromes such as severe aplastic anemia. The strongest predictor of progression and death from invasive mold infection in the cancer/ HSCT setting is the duration of neutropenia. Any modality which increases the granulocyte count during periods of profound neutropenia and severe infection is thus likely to be of clinical benefit. In the 1970-80 s, collection of granulocyte concentrates by apheresis of healthy donors stimulated with corticosteroids alone yielded products with an insufficient number of granulocytes to substantially raise the circulating counts in neutropenic patients. Transfusion of such components was variably associated with clinical benefit. More recently, the ability to give donors recombinant human granulocyte colony-stimulating factor (G-CSF) in combination with corticosteroids (dexamethasone) dramatically increases the circulating neutrophil count prior to apheresis and results in the collection of granulocyte concentrates containing 2 to 6 times as many cells as those collected using steroids alone. Transfusion of granulocyte concentrates collected after G-CSF and dexamethasone stimulation of the donor typically increases the recipient s granulocyte count by 1,000 cells/uL, and the increase in counts is generally sustained for 24 to 48 hours. Transfusion of daily or every other day granulocytes derived by apheresis of G-CSF and dexamethasone-stimulated donors has been associated in observational and retrospective studies with clearance of life-threatening infections in neutropenic patients, but a single small randomized prospective study did not demonstrate improved survival in neutropenic infected patients who received granulocytes. Granulocyte components are not recognized as a licensed blood component by the Food and Drug Administration (FDA), and neither G-CSF nor dexamethasone is approved by the FDA for use in allogeneic granulocytapheresis donors. Studies at the NIH Department of Transfusion Medicine (DTM) have defined the optimal timing and dose of these drugs in granulocyte donors, and these components have been used for clinical care since 1996. Short term adverse effects of G-CSF and dexamethasone, including bone pain, myalgia, headache, insomnia and fatigue, are well known and possible long-term effects, including cataracts from serial steroid administration, have been described. The purpose of the current protocol is to determine the operational feasibility of managing a volunteer community donor granulocytapheresis program and to provide informed consent for the administration of filgrastim and dexamethasone to volunteer donors donating granulocytes by apheresis. Donor accrual and retention, immediate short term adverse effects of G-CSF and dexamethasone, and any long-term effects, will be assessed in healthy subjects who will be permitted to donate granulocytes a maximum of 12 times per year. Reasonable efforts will be made to equitably distribute opportunities for granulocyte donation so that the maximal number of annual donations is not met by any one donor.Participants will be selected based on general blood donor eligibility criteria, adequacy of antecubital venous access, and interest in the program. Most subjects will already have experience as plateletpheresis donors. The toxicity of granulocyte transfusions and the survival and discharge rates of the transfusion recipients will be monitored, but the protocol is not designed to evaluate the efficacy of granulocyte transfusions.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Donors shall meet all donor eligibility criteria for allogeneic blood donors, as defined in the most recent editions of the AABB Standards and FDA Code of Federal Regulations (21CFR640). In addition, donors shall meet the following restrictions:
* Age greater than or equal to18 and less than or equal to 75 years
* If hypertension is present, must be well-controlled on medications
* If peptic ulcer disease has been diagnosed in the past, symptoms must be well-controlled on medications
* If cataracts have been diagnosed in the past, records from subject s ophthalmologist must be obtained indicating type of cataract. If PSC was diagnosed in the past, subject may receive G-CSF but not dexamethasone. The only exception to this is a history of bilateral cataract extractions due to PSC.

EXCLUSION CRITERIA:

* Information obtained from health history screen that does not meet the allogeneic donor eligibility criteria of the AABB Standards or the FDA CFR.
* Weight less than 50 kg (110 lbs).
* History of coronary heart disease
* Uncontrolled hypertension (systolic BP >160, diastolic BP >100)
* Diabetes mellitus requiring insulin
* Active, symptomatic peptic ulcer disease
* History of iritis or episcleritis
* Sickle cell disease (sickle trait is acceptable). Testing for hemoglobin S is not required.
* Lithium therapy
* Pregnancy or nursing (breast feeding)
* Renal function eGFR < 45 ml/min/1.73m(2)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2012-12-31 (Actual); Primary Completion 2032-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Operational feasibility and impact of managing a volunteer community donor granulocytapheresis program | Annually
  Establishment of a donor registry sufficient to meet the granulocyte transfusion needs of all Clinical Center patients. This endpoint shall include(1) the number of donors recruited into the program (2) the retention rate of donors in the program, assessed by number of donations per year per donor, cumulative number of granulocyte donations per donor, and duration of participation in the program per donor (3) the number of requests for a course of granulocytes per year and the number and percent of these requests that could be met, including the percent of all requested transfusion days on which granulocytes were available (4) the impediments to meeting all requests for granulocyte components, with an analysis of whether these are due to lack of an adequate donor supply or lack of adequate staffing or apheresis capacity (5) characteristics of the patients who are supported by a course of granulocyte transfusions.

SECONDARY OUTCOMES:
Long-term adverse effects of repeated doses of filgrastim and dexamethasone in volunteer apheresis donors | Annually
  Changes in CBC or health histories over time in donors continuing in the program.
Frequency and severity (symptom grade) of acute adverse effects due to a single dose of filgrastim and dexamethasone in volunteer donors | Annually
  Frequency and severity of acute adverse events related to G-CSF and dexamethasone in granulocyte donors.

CONTACTS AND LOCATIONS:
Overall Officials: Kamille A West-Mitchell, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Wingard JR, Carter SL, Walsh TJ, Kurtzberg J, Small TN, Baden LR, Gersten ID, Mendizabal AM, Leather HL, Confer DL, Maziarz RT, Stadtmauer EA, Bolanos-Meade J, Brown J, Dipersio JF, Boeckh M, Marr KA; Blood and Marrow Transplant Clinical Trials Network. Randomized, double-blind trial of fluconazole versus voriconazole for prevention of invasive fungal infection after allogeneic hematopoietic cell transplantation. Blood. 2010 Dec 9;116(24):5111-8. doi: 10.1182/blood-2010-02-268151. Epub 2010 Sep 8. PMID 20826719
- [Background] Baddley JW, Andes DR, Marr KA, Kontoyiannis DP, Alexander BD, Kauffman CA, Oster RA, Anaissie EJ, Walsh TJ, Schuster MG, Wingard JR, Patterson TF, Ito JI, Williams OD, Chiller T, Pappas PG. Factors associated with mortality in transplant patients with invasive aspergillosis. Clin Infect Dis. 2010 Jun 15;50(12):1559-67. doi: 10.1086/652768. PMID 20450350
- [Background] Stroncek DF, Yau YY, Oblitas J, Leitman SF. Administration of G--CSF plus dexamethasone produces greater granulocyte concentrate yields while causing no more donor toxicity than G--CSF alone. Transfusion. 2001 Aug;41(8):1037-44. doi: 10.1046/j.1537-2995.2001.41081037.x. PMID 11493736
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2012-CC-0096.html